CLINICAL TRIAL: NCT06323044
Title: MedSupport: A Novel Multilevel Intervention to Identify and Address Barriers to Pediatric Medication Adherence
Brief Title: MedSupport Intervention to Identify and Address Barriers to Pediatric Medication Adherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I-3920723; NCI-2024-01734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I-3920723 (Other: Roswell Park Cancer Institute); R01CA283501 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (MedSupport) (Experimental): Participants receive the MedSupport intervention consisting of three components: universal screening for adherence barriers, tailored virtual education enhancement, and communication of barriers to activate multidisciplinary healthcare teams for 12 months. Participants also use the MEMS device to track oral chemotherapy adherence at baseline and follow-up. Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Survey Administration
- Arm B (usual care) (Active Comparator): Participants receive usual care consisting of medical consultations and supportive care for 12 months. Participants also use the MEMS device to track oral chemotherapy adherence at baseline and follow-up. Patients also undergo blood sample collection throughout the study.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Interview; Other: Medical Device Usage and Evaluation; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm B (usual care)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Electronic Health Record Review — Ancillary studies
Other: Interview — Ancillary studies
Other: Medical Device Usage and Evaluation — Receive MedSupport intervention
  Arms: Arm A (MedSupport)
Other: Medical Device Usage and Evaluation — Use MEMS device
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial identifies and addresses barriers to pediatric medication adherence among families of children with acute lymphoblastic leukemia. Pediatric nonadherence (noncompliance) to medication is a significant public health problem, and rigorous research repeatedly documents that nonadherence increases risk for hospitalization, healthcare cost, disease progression, and death. Pediatric acute lymphoblastic leukemia (ALL) patients who miss 5% of 6-mercaptopurine (6-MP) doses within the 2-year 6-MP regimen have a 2.7-fold risk of cancer that comes back after a period of improvement (relapse). To address these families' needs, researchers have developed MedSupport, a theory-based multilevel intervention with targets at the organizational, healthcare team, and caregiver levels that is designed to address root barriers to medication adherence. This study is being done to better understand families' experiences giving their child oral chemotherapy at home and to help families cope with the day-to-day challenges of giving their child medication.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the proportion of pediatric ALL patients with 6-mercaptopurine (6-MP) chemotherapy adherence 95% or higher based on Medication Event Monitoring System (MEMS) data collected during the Consolidation II (1st year of therapy) and Continuation (2nd year of therapy) treatment phases in patients randomized to either MedSupport intervention or usual care.

EXPLORATORY OBJECTIVES:

I. To compare the proportion of pediatric acute lymphoblastic leukemia (ALL) patients with 6-mercaptopurine chemotherapy adherence based on 6-MP metabolite analysis of peripheral blood biospecimens collected during the Consolidation II and Continuation phases of treatment in patients randomized to either MedSupport intervention or usual care. (PATIENT) II. To use statistical modeling to examine potential mechanisms/mediators (medication barriers verse [vs.] social support, medication beliefs) of intervention efficacy in patients randomized to either MedSupport intervention or usual care. (PATIENT) III. To use statistical modeling to explore potential moderators of intervention efficacy including child age, caregiver socioeconomic status, race, ethnicity, and household structure in patients randomized to either MedSupport intervention or usual care. (PATIENT) IV. To determine parent intervention uptake by examining engagement with the screening questionnaire among parents from the intervention arm as a percentage based upon the ratio of the number of screening questionnaires completed to the number of questionnaires the participant was eligible to complete. (CAREGIVER) V. To assess whether parents from the intervention arm engaged with the educational videos as a percentage based upon the ratio of the number of minutes of videos watched compared to the number of minutes of educational videos the participant was prompted to view. (CAREGIVER) VI. To examine the strategies that may hinder or support implementation within routine care by assessing how parents from the intervention arm rated the acceptability, appropriateness, and feasibility of the MedSupport intervention. (CAREGIVER) VII. To explore barriers and facilitators to adoption, feasibility, and sustainability of the MedSupport intervention by examining the responses of a sample of 20 parent participants from the intervention arm who participate in semi-structured qualitative interviews. (CAREGIVER) VIII. To determine healthcare provider uptake by examining documentation of 4 weeks of adherence/medication-related consultations from intervention arm patient's Electronic Health Record (EHR) following a medication barrier alert. (INSTITUTIONAL) IX. To examine strategies that may hinder or support implementation within routine care by assessing healthcare provider ratings of the acceptability, appropriateness, and feasibility of the MedSupport intervention. (INSTITUTIONAL) X. To explore barriers and facilitators to adoption, feasibility, implementation, organizational/contextual factors that support maintenance and cost of the MedSupport intervention by examining the responses of a sample of 20 healthcare providers who participated in semi-structured qualitative interviews. (INSTITUTIONAL)

OUTLINE: Participants are randomized to 1 of 2 groups.

GROUP A: Participants receive the MedSupport intervention consisting of three components: universal screening for adherence barriers, tailored virtual education enhancement, and communication of barriers to activate multidisciplinary healthcare teams for 12 months. Participants also use the MEMS device to track oral chemotherapy adherence at baseline and follow-up. Patients also undergo blood sample collection throughout the study.

GROUP B: Participants receive usual care consisting of medical consultations and supportive care for 12 months. Participants also use the MEMS device to track oral chemotherapy adherence at baseline and follow-up. Patients also undergo blood sample collection throughout the study.

After completion of study intervention, participants are followed up at 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child who is diagnosed and receiving first line therapy for acute lymphoblastic leukemia (ALL) at a study site.
* Parent's child patient is age 365 days to < 19 years at time of study entry.
* Parent's child patient's therapy must include 6-mercaptopurine (6-MP) administered orally or by nasogastric (NG) tube.
* Parent has verbal English, French, or Spanish fluency.
* Parent has a smartphone or access to a computer with an Internet connection.
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.

Exclusion Criteria:

* Parent is unwilling or unable to follow protocol requirements.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | Up to 1 year
  Will be summarized by timepoint (baseline, 6-months, and 1-year) and condition using descriptive statistics and graphical summaries. The primary analysis will model log adherence as a function of condition, timepoint, their two-way interaction, and random family (accounting for the longitudinal measures within a family unit) and site (accounting for between cancer center variability) effects using a linear mixed model (LMM). Bonferroni adjusted tests about the appropriate contrasts of model estimates will be used to compare: 1) the mean change in adherence within each condition, 2) retention of effect at 12-months within each condition, and 3) the mean change in adherence between conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Kara M Kelly, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States